CLINICAL TRIAL: NCT00508729
Title: Effect of Traditional Chinese Medicine on Gastrointestinal Function Recovery and Nutrition Support in Severe Acute Pancreatitis
Brief Title: Effect of Traditional Chinese Medicine on GI Function Recovery and Nutrition Support in SAP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Collaborators: Peking Union Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006BAI04A15-1
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Pancreatitis, Acute Necrotizing
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Qingyi granules

SUMMARY:
With multicenter randomized control clinical evaluation investigations, the effect of traditional Chinese medicine on gastrointestinal function recovery and nutrition support in early stage of severe acute pancreatitis (SAP) was evaluated, and the therapeutic effects, safety and indications assured. Drawing in latest research fruits at home and abroad, a clinical practical guideline would be formed, to be popularized all over China.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 yr-70 yr
* Complying with the diagnostic standard of acute pancretitis (clinical symptoms and signs, elevated blood and urine amylase, and imaging criteria)
* Conforming to 3 or more Ranson's criteria and APACHE-II score larger than 8, Balhazar CT score larger than 5

Exclusion Criteria:

* Pregnancy
* Nursing mother
* Critical cases of advanced tumor
* On the verge of death (estimated to be moral in 12h)
* Severe visceral function disturbance
* Patients undergoing other therapeutic research that might interfere with the present study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-10; Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | endpoint of the trial
Morbidity | endpoint of the trial
Hospitalization days | endpoint of the trial
Total expenses | endpoint of the trial

SECONDARY OUTCOMES:
G-I tract function: nature of abdominal pain, intra-abdominal pressure, number of bowel movements | The above criteria should be tested on admission, and 24h, 48h and 72h later, 5d, 7d, and 2wks after admission, and on the day of discharge
Parameters of nutrition | The above criteria should be tested on admission, and 24h, 48h and 72h later, 5d, 7d, and 2wks after admission, and on the day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Naiqiang Cui, Dr, Principal Investigator — Tianjin Nankai Hospital; Zhuming Jiang, Dr, Principal Investigator — Peking Union Medical College Hospital
Locations (10):
- China (10):
  - Affiliated Hospital of Guangdong Medical College, Zhanjiang, Guangdong
  - Guizhou Province People's Hospital, Guiyang, Guizhou
  - The 1st Affiliated Hospital, Dalian Medical Unversity, Dalian, Liaoning
  - West China Hospital, Sichuan Unversity, Chengdu, Sichuan
  - Zhejiang Province People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Province Traditional Chinese Medicine Hospital, Hangzhou, Zhejiang
  - Dongzhimen Hospital of Beijing Traditional Chinese Medicine University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Longhua Hospital of Shanghai Traditional Chinese Medicine Unversity, Shanghai
  - Tianjin Nankai Hospital, Tianjin